CLINICAL TRIAL: NCT01502722
Title: Effect of Ingestion of Sugary Drinks on Thirst Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Pedro Miguel Fernandes Ramos de Carvalho, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IHS/FCNAUP-001
Record Dates: First submitted 2011-11-22; First posted 2012-01-02 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Thirst

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 - Crossover (Experimental): This group will drink water in the 1st study.
  Interventions: Behavioral: Effect of ingestion sugary and sweetened drinks on thirst
- Group 2 - Crossover (Experimental): This group will drink Pineapple Soda in the 1st study
  Interventions: Behavioral: Effect of ingestion sugary and sweetened drinks on thirst
- Group 3 - Crossover (Experimental): This group will drink Pineapple Diet Soda in the 3rd study
  Interventions: Behavioral: Effect of ingestion sugary and sweetened drinks on thirst

INTERVENTIONS:
Behavioral: Effect of ingestion sugary and sweetened drinks on thirst — The participants will drink Water (control group), Decarbonized Pineapple Soda (11% sugar)and Decarbonized Pineapple Diet Soda (1% Sugar and Sucralose). The beverages will be presented chilled but without ice in 500 ml portions in opaque plastic containers and participants will be asked to consume the entire amount within 15 min. The beverages will be tested previously in laboratory in order to obtain their pH and osmolality.
  Other Names: Effect of ingestion of water, soda and diet soda on thirst; Diferences between sweeteners and sugar on thirst

SUMMARY:
The purpose of this study is to determine if regular soft drinks (with sugar) have the same effect on thirst as diet soft drinks(with sweeteners).

DETAILED DESCRIPTION:
Participants should be in the laboratory at 8.00 in order to collect the values of weight, height, total body water, intracellular water and extracellular water in a Segmental Multi Frequency Body Composition Monitor (TANITA MC 180 MA®). Then, a blood sample will be collected for analysis of blood glucose and osmolality. They will sit at individual tables for the duration of the session and were allowed to read, listen to music with earphones, or use their portable computers with the exception of internet access to minimize visual cues (e.g., unwanted publicity for beverages or visiting Web sites showing pictures of food and drinks), which may have effect on thirst. Breakfast will be served at 9.30 on every occasion and preload stimuli will be offered exactly 60 minutes after breakfast (at 10.30). Lunch will be provided at 13.00. Motivational ratings will be first obtained at the end of collection of blood sample (baseline or time 0) and every 30 minutes thereafter until the lunch time (times 1 through 7). After lunch (time 8), participants will complete the last set of ratings and will bring a food diary to record all food and fluid intake until 00.00 that day.

ELIGIBILITY:
Inclusion Criteria:

* body mass index(BMI) between (18,5 - 25 kg/m2)
* regular consumers of breakfast
* stable in weight for the past 6 months
* not dieting to gain or lose weight
* like all drinks and food available in study

Exclusion Criteria:

* pregnant and nursing women
* smokers
* athletes
* subjects under medication(except oral contraceptives in women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Motivational Ratings | 1 day
  Participants will rate their hunger, thirst, nausea, mouth dryness, desire to eat, desire to drink using nine point category scales. The unipolar adjective scales were anchored at each end with labels: 1 = not at all and 9 = extremely. Participants also rated their liking for the beverage along nine point hedonic preference scales where 1 = dislike extremely and 9 = like extremely

SECONDARY OUTCOMES:
Food Behavior After Intervention | 1 day
  After lunch, participants will bring a food diary to record all food and fluid intake until 00.00 that day. Then, we will analyse total calories ingested, total fluid ingested and the volume of sugar and sugary beverages ingested.
Amount of water ingested | 1 day
  After the ingestion of 3 preloads with the beverages in study (water, pineapple soda and pineapple diet soda), the participants will lunch the same meal bu the water ingestion will be ad libitum.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro R Carvalho, PhD Student, Principal Investigator — Faculdade de Ciências da Nutrição e Alimentação - Universidade do Porto; Vitor H Teixeira, PhD, Study Director — Faculdade de Ciências da Nutrição e Alimentação - Universidade do Porto
Locations (1):
- Faculdade de Ciências da Nutrição e Alimentação da Universidade do Porto, Porto, Porto District, Portugal

REFERENCES:
- [Background] Monsivais P, Perrigue MM, Drewnowski A. Sugars and satiety: does the type of sweetener make a difference? Am J Clin Nutr. 2007 Jul;86(1):116-23. doi: 10.1093/ajcn/86.1.116. PMID 17616770
- [Background] Almiron-Roig E, Drewnowski A. Hunger, thirst, and energy intakes following consumption of caloric beverages. Physiol Behav. 2003 Sep;79(4-5):767-73. doi: 10.1016/s0031-9384(03)00212-9. PMID 12954421